CLINICAL TRIAL: NCT05272839
Title: Association Between Natural Hypoglycemic Foods and Blood Sugar Level: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Antenna Foundation (Other)
Collaborators: Khon Kaen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiabetesThai22
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: At the first visit, patients will be randomly assigned to control group or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoglycemic food group (Experimental): The patient will choose 2 food products clinically validated against diabetes, at the same dosage and the same mode of preparation as in the reference clinical trials. This will be done additionally to healthcare advice and standard medication if any.
  Interventions: Dietary Supplement: Hypoglycemic food group
- Control group (Placebo Comparator): The control group will receive only dietary advice and standard medication if any.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Hypoglycemic food group — A booklet with 4 common food products, clinically validated against diabetes, with instructions for use will be presented to the diabetic patient. The selected food products have been assessed as anti-diabetic for humans through at least one fair randomized comparative clinical trial, with a follow-up of several weeks or months. While continuing to take his/her standard medication if any, the patient will be encouraged to follow his/her preferences within the established list of foods and spices: he is expected to choose 2 plants from the list and to consume each of them every day during the whole duration of the trial (12weeks).
  Arms: Hypoglycemic food group
Dietary Supplement: Control group — The control group will receive only lifestyle and dietary recommendations.
  Arms: Control group

SUMMARY:
Type 2 diabetes patients often do not reach desired control of glycemia despite guidance on changing lifestyle and diet as well as the use of conventional anti-diabetic medication. Parallely in recent years, an array of comparative clinical studies have demonstrated the anti-diabetic effect of more than 10 common spices and food products. Objectives: to evaluate whether proposing a choice of spices and foods products with hypoglycemic effect to diabetic patients can help better control diabetes.

DETAILED DESCRIPTION:
Diabetic type II patients would be encouraged to eat what they like within a list of food products with hypoglycemic effect, at a similar dosage and preparation mode than the one in the reference clinical trials.

This pilot project will be conducted as a randomized controlled trial with 2 arms over 12 weeks: 1. training patients about hypoglycemic spices and foods alongside their usual anti-diabetic treatment, versus usual anti-diabetic treatment alone.

Expected results: Confirmation of the hypothesis that daily consuming spices and foods with hypoglycemic effect to diabetic patients can help better control diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with poorly controlled glycemia, i.e. at least one of the following measurements:

  1. Fasting plasma glucose (FPG) values ≥ 7.0 mmol/L (126 mg/dl), or 2-h post-load plasma glucose ≥ 11.1 mmol/L (200 mg/dl), or HbA1c > 6.5% (48 mmol/mol); or a random blood glucose ≥ 11.1 mmol/L (200 mg/ dl), despite ≥ 3 months usual care (lifestyle + medication if applicable).

Exclusion criteria:

1. Severe and unstable complications of diabetes: end-organ damage such as nephropathy, retinopathy, neuropathy, etc...
2. Patients with rapid insulin,
3. Any health condition that requires urgent attention,
4. Patients with a cognitive or sensory impairment that may prevent conducting the interview,
5. HbA1c > 11.5%
6. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Decrease of ≥ 0.5mmol/L in FPG | 12 weeks
  Percentage of patients in each group reaching a decrease of ≥ 0.5mmol/L in FPG over 12 weeks
Decrease of ≥ 0.5 points of percentage of HbA1c | 12 weeks
  Percentage of patients in each group reaching a decrease of ≥ 0.5 points of percentage from the baseline value in HbA1c over 12 weeks

SECONDARY OUTCOMES:
Mean change of FPG | 12 weeks
  Mean change of FPG e.g. differences between baseline values and values at 12 weeks
Target glycemia | 12 weeks
  Proportion of patients in each group reaching target glycemia over 12 weeks
Weight | 12 weeks
  Mean change of weight [kg] over 12 weeks
Mean change of HbA1c | 12 weeks
  Mean change of HbA1c e.g. differences between baseline values and values at 12 weeks
Blood pressure | 12 weeks
  Mean change of systolic and diastolic blood pressure [mmHg] over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Graz, MD, MPH, Study Director — Antenna Foundation

IPD SHARING:
Plan to Share IPD: Yes
IPD will be kept in a safe location in Khon Kaen University hospital. It will be available in an anonymous manner upon request and after deidentification.
Supporting Information: Study Protocol
Time Frame: April 2023 up to April 2033
Access Criteria: It will be accessible to any researchers or reviewers who might review the data and perhaps perform some new data analysis. The decision will be in the hands of the Principal investigator and colleagues in Khon Kaen University, plus health and ethical authorities following legislation.

REFERENCES:
- [Background] Willcox ML, Elugbaju C, Al-Anbaki M, Lown M, Graz B. Effectiveness of Medicinal Plants for Glycaemic Control in Type 2 Diabetes: An Overview of Meta-Analyses of Clinical Trials. Front Pharmacol. 2021 Nov 26;12:777561. doi: 10.3389/fphar.2021.777561. eCollection 2021. PMID 34899340